CLINICAL TRIAL: NCT07274111
Title: Virtual Reality to Manage Pediatric Gastrointestinal Endoscope-related Anxiety, Post Procedural Pain, and Recovery Time: A Randomized Control Trial
Brief Title: Virtual Reality as a Nursing Intervention for Anxiety and Pain in Pediatric Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Rasha Gad, Lecturer of pediatric Nursing, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0493
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2023-06

CONDITIONS: Gastrointestinal Endoscopy; Procedural Anxiety; Pain
Keywords: Pediatric Nursing; Virtual Reality (VR); Pediatric Endoscopy; Anxiety; Pain
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind randomized controlled trial. Participants and clinical staff were aware of group allocation due to the visible nature of the VR intervention. However, the statistician analyzing the data was blinded to group assignments to minimize assessment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) Intervention (Experimental): Participants in this arm received a one-minute immersive Virtual Reality (VR) session prior to gastrointestinal endoscopy. Using a head-mounted display with age-appropriate preloaded environments (roller coaster, space, wildlife, travel scenes), the nurse assisted in headset fitting and adjustment. The VR session aimed to reduce pre-procedural anxiety and enhance comfort. All assessments and procedures were conducted following the same standardized schedule as the control group to ensure comparability.
  Interventions: Behavioral: Virtual Reality Head-Mounted Display
- Standard Care (Control) (No Intervention): Participants in this arm received standard pre-procedural care without exposure to Virtual Reality. The usual preparation and education were provided by the endoscopist, anesthesiologist, and nurse according to hospital policy. Children underwent identical assessment points as the intervention group, including evaluation of anxiety, physiological stability, pain, and recovery time, to allow valid comparison between groups under consistent clinical conditions.

INTERVENTIONS:
Behavioral: Virtual Reality Head-Mounted Display — Children assigned to the experimental arm received a one-minute immersive session using a virtual reality head-mounted display before gastrointestinal endoscopy. The device contained age-appropriate preloaded applications featuring realistic visual and auditory environments, such as roller coasters, space exploration, wildlife parks, and travel scenes. The nurse assisted each child in properly fitting and adjusting the headset to ensure comfort and clarity. The VR session was administered immediately before transfer to the endoscopy room to reduce pre-procedural anxiety and enhance relaxation.
  Other Names: Immersive VR Session
  Arms: Virtual Reality (VR) Intervention

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of a virtual reality (VR) intervention in managing anxiety, post-procedural pain, and recovery time among pediatric patients undergoing gastrointestinal (GI) endoscopy. The study is conducted at the Pediatric Gastrointestinal Endoscopy Unit, Mansoura University Children's Hospital, Egypt. Eligible children are randomly assigned to either a VR intervention group or a control group receiving standard care. The VR group uses a head-mounted display featuring age-appropriate immersive applications before endoscopy. Measured outcomes include anxiety levels, physiological stability, post-procedural pain, and recovery duration. The study follows CONSORT guidelines and ethical principles outlined in the Declaration of Helsinki.

DETAILED DESCRIPTION:
This prospective randomized controlled experimental study investigates the use of virtual reality (VR) as a non-pharmacological nursing intervention to reduce anxiety and enhance recovery outcomes in pediatric patients undergoing gastrointestinal endoscopic procedures. The study is conducted at the Pediatric Gastrointestinal Endoscopy Unit of Mansoura University Children's Hospital, located in Mansoura City, Dakahlia Governorate, Egypt.

Participants include children aged 6-15 years scheduled for their first GI endoscopy who demonstrate an interest in technology and consent to participate. Children with seizure disorders, cardiac diseases, visual or hearing impairments, developmental delays, motion sickness, or those undergoing chemotherapy are excluded.

Following ethical approval and informed consent, participants are randomly allocated in a 1:1 ratio to either the VR intervention or control group. Both groups receive a standardized pre-procedural education session delivered by the endoscopist, anesthesiologist, and nurse. In the waiting area, baseline assessments include demographic characteristics, state and trait anxiety (using the State-Trait Anxiety Inventory for Children), physiological parameters (respiratory rate, heart rate, and oxygen saturation), and pain level (using the Wong-Baker FACES Pain Rating Scale).

Children in the VR group wear a head-mounted display containing preloaded age-appropriate immersive environments, such as virtual roller coasters, space exploration, wildlife parks, and travel scenes, for one minute before entering the endoscopy room. The nurse assists with headset adjustment and ensures proper device hygiene. The control group receives standard pre-procedural care without VR exposure.

Anxiety and physiological indicators are reassessed in the endoscopy room prior to anesthesia induction. Post-procedural pain and recovery duration (time spent in the recovery room until discharge) are recorded afterward. Data are analyzed using SPSS version 26, employing descriptive statistics, independent t-tests, chi-square tests, and non-parametric alternatives where appropriate. Statistical significance is set at p < .05.

This trial aligns with CONSORT reporting standards and aims to provide evidence on the clinical value of VR as an effective, child-friendly nursing intervention for anxiety and pain management in pediatric endoscopy settings.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-15 years scheduled to undergo a gastrointestinal endoscopic procedure.
* First-time endoscopy patients (no prior endoscopic experience).
* Willing to participate, with informed consent from parents/guardians and child assent.

Interest in technology and ability to tolerate a brief VR experience.

- Physically and cognitively able to complete the anxiety and pain assessment tools (STAI-CH and FACES scales).

Exclusion Criteria:

* Children with a known history of seizure disorders or cardiac diseases.
* Presence of active infection, burns, or trauma involving the periorbital skin, eyes, nasal bridge, external ear, scalp, or hair.
* Visual or hearing impairments that would interfere with VR use.
* Developmental delays (including autism spectrum disorders) that significantly limit cooperation or understanding of instructions.
* Active psychosis or symptoms of intoxication.
* History of severe motion sickness.
* Children currently undergoing chemotherapy.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Children's Anxiety Levels | Trait subscale was assessed only prior to the child's entry while the State subscale was assessed prior to entrance into the endoscopy room (pre-procedure) and before the induction of anesthesia (peri-procedure).
  Anxiety levels was measured using the State-Trait Anxiety Inventory for Children (STAI-CH). Both the trait and state subscales was used. The primary outcome was the difference in state anxiety scores before and during the intervention between the VR and control groups. Each item is scored on a 3-point Likert scale, with total scores ranging from 20 to 60, where higher scores indicate greater anxiety.
Change in Pain Level | Two time points: pre-procedural pain level (immediately before entering the endoscopy room) and post-procedural pain level (30 minutes post-procedure in the recovery unit).
  pain will be measured using the Wong-Baker FACES Pain Rating Scale, which ranges from 0 (no pain) to 10 (worst pain). The outcome represents the mean difference in pain levels between the VR and control groups following the endoscopic procedure.
Recovery Duration | Measured from the time of entry into the recovery room until discharge, assessed up to 300 minutes.
  Recovery time will be measured as the total duration of each child's stay in the recovery room (recorded in minutes and presented in hours) from entry into the recovery unit until discharge criteria are met. The outcome represents the mean recovery duration between the VR and control groups.

SECONDARY OUTCOMES:
Change in respiratory rate | Respiratory rate was assessed immediately before entering the endoscopy room (pre-procedure) and again prior to anesthesia induction (peri-procedure).
  Respiratory rate was recorded in breaths per minute (bpm) using the bedside multiparameter monitor. The outcome reflects the mean change in respiratory rate between baseline and the peri-procedural time point.
Change in heart rate | Heart rate was assessed prior to entrance into the endoscopy room (pre-procedure) and before the induction of anesthesia (peri-procedure).
  Heart rate was recorded in beats per minute using the bedside multiparameter monitor. The outcome reflects the mean change in heart rate between baseline and the peri-procedural time point.
Change in Oxygen Saturation | Oxygen saturation was assessed prior to entrance into the endoscopy room (pre-procedure) and before the induction of anesthesia (peri-procedure).
  Oxygen saturation was measured using the bedside multiparameter monitor and expressed as a percentage (SpO₂). The outcome reflects the mean change in oxygen saturation between baseline and the peri-procedural time point.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Gad, Ph.D, Principal Investigator — Mansoura University, Faculty of Nursing
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No